CLINICAL TRIAL: NCT00560469
Title: Impaired Adipogenesis in Insulin Resistance: Pilot Clinical and In Vitro Studies
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Richard Pratley, MD, University of Vermont
Other Study IDs: R21DK080386 (NIH); R21DK080386 (NIH); 1R21DK80386-1; 958
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2010-09

CONDITIONS: Adipocyte Differentiation; Insulin Resistance
Keywords: Adipokines; Inflammation; Metabolic syndrome
MeSH Terms: conditions — Insulin Resistance; Inflammation; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Adipose tissue, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Men and Women over age 40 who are obese (BMI>30) and insulin-resistant.
  Interventions: Other: Administration of 70% deuterated water
- 2: Men and women over age 40 who are obese (BMI>30) and insulin-sensitive.
  Interventions: Other: Administration of 70% deuterated water

INTERVENTIONS:
Other: Administration of 70% deuterated water — Subjects will drink 70% deuterated water daily for 8 weeks.

SUMMARY:
Obesity is a strong risk factor for developing type 2 diabetes (T2DM), but the reasons for this are not fully understood. In particular, it is not known why some obese people develop T2DM while other obese individuals do not. This study tests whether differences in fat cells (adipocytes) are to blame. Even in adults, fat cells are constantly being formed to replace old fat cells and to respond to the body's need to store excess energy. The ability to form new fat cells may be diminished in some individuals, leading to larger fat cells. These large fat cells secrete hormones that may increase risk for T2DM. This study tests whether fat cells from obese insulin resistant subjects (who are at risk for developing T2DM) form at a slower rate than those from insulin sensitive subjects (who are at lower risk for developing T2DM).

To address this question we will recruit and study two groups of obese subjects, selected to be similar in age, gender and degree of obesity. One group of subjects will be obese and insulin resistant (the OIR group), while the other will be comparably obese, but insulin sensitive (OIS). Subjects will undergo a series of studies to characterize their metabolism including measurement of body fat by DEXA scanning, oral glucose tolerance (a test used to diagnose diabetes) and measurement of insulin sensitivity in response to an infusion of insulin (a research study used to classify patients into the OIR and OIS groups). Small samples of fat (from just under the skin of the belly and the buttocks) will obtained using a needle on two occasions over 12 weeks. During these 12 weeks, subjects will drink a small amount of water that contains a non-radioactive label. This labeled water will allow us to measure the rate of growth of new fat cells in the body. We will also look at the rate of growth of fat cells obtained from these biopsies in the laboratory.

The results of this study may tell us more about why certain obese people develop diabetes and why others do not. This might lead to new ways to prevent or treat T2DM.

DETAILED DESCRIPTION:
Overview of design: To address the specific aims of this study we will recruit and study two groups of obese subjects, selected to be similar in age, gender and BMI. Based on the results of an oral glucose tolerance test (OGTT) and hyperinsulinemic-glucose clamp, one group will be obese and insulin resistant (OIR) and one will be obese and insulin sensitive (OIS). Subjects will undergo measurement of body fat and fat distribution, oral glucose tolerance, in vivo insulin sensitivity, percutaneous needle biopsies of subcutaneous abdominal and gluteal fat and in vivo measurement of SVC and adipocyte turnover using the D2O DNA labeling technique. Adipocyte size and the expression of pro-inflammatory cytokines and adipokines will be compared in the two groups. Primary cultures of preadipocytes will be derived from subjects and proliferation and differentiation measured in vitro and compared to in vivo measures.

Measurement of adipocyte proliferation and differentiation in vivo: The stable isotope technique of Hellerstein et al. for the measurement of slowly dividing cells is based on the incorporation of deuterium oxide (D2O) into DNA. This method has been used to estimate rates of turnover of adipocytes and stromal vascular cells in healthy normal volunteers. It has not, to date, been employed to compare groups of subjects who may differ in their adipogenic propensity. A major objective of the study, therefore, is to evaluate the utility of this approach for quantifying in vivo differences in adipocyte and SVC turnover between groups that vary by insulin sensitivity and to compare the in vivo measures obtained using this technique with in vitro measures of adipogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 40-65 who are obese (BMI>30)and weight stable for 6 months prior to enrollment.

Exclusion Criteria:

* Acute or chronic medical conditions that would contraindicate participation in the research testing
* Pregnant or nursing women
* HbA1c>6.5%
* Active alcohol or drug abuse
* Weight >300 pounds.
* Smoking

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
In vitro rates of adipocyte turnover | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Pratley, MD, Principal Investigator — University of Vermont
Locations (1):
- Fletcher Allen Health Care, South Burlington, Vermont, United States